CLINICAL TRIAL: NCT04904081
Title: The Use of Indocyanine Green Angiography in Pediatric Colorectal Surgery: A Feasibility Randomized Controlled Trial
Brief Title: Feasibility of Use of Indocyanine Green in Pediatric Colorectal Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #202103
Record Dates: First submitted 2021-05-14; First posted 2021-05-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Hirschsprung Disease; Anorectal Malformations
MeSH Terms: conditions — Hirschsprung Disease; Anorectal Malformations | interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind (participants only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Indocyanine Green [ICG]) (Experimental): The ICG group will involve the patient receiving standard care for either HD or ARM, in addition to 1.25mg (maximum dose less than 2mg/kg body weight) of ICG intraoperatively, administered intravenously. ICG will be administered by a member of the anesthesia team when directed by the surgeon (research team member).
  Interventions: Drug: Indocyanine green
- Control Arm (Standard Care) (No Intervention): The Standard Care group will have no change to the medical and surgical care they receive while in the hospital. The surgeon will perform the surgery as they normally would outside of this study. This involves a laparoscopic-assisted transanal pullthrough surgery.

INTERVENTIONS:
Drug: Indocyanine green — The ICG group will involve the patient receiving standard care for either HD or ARM, in addition to 1.25mg (maximum dose less than 2mg/kg body weight) of ICG intraoperatively, administered intravenously. ICG will be administered by a member of the anesthesia team when directed by the surgeon (research team member).
  Arms: Treatment Arm (Indocyanine Green [ICG])

SUMMARY:
Hirschsprung's Disease (HD) and anorectal malformations (ARM) are both paediatric diseases of the colon and rectum. Both of these conditions require surgery in order to correct them, frequently needing sections of the bowel to be removed. Some complications of removing parts of the bowel include forming a stricture (a narrowing of the place where the bowel is reattached), and leak from the join. These can be devastating complications, and can significantly impact a patient's quality of life. Indocyanine green (ICG) is a medication that binds to blood vessels and can be visualized using special cameras in the operating room. Once it binds, it "lights up" green on this equipment. This lends the advantage of being able to better see which parts of the bowel get good blood flow. The theory is that good blood flow can reduce the risks of previously mentioned complications. This has been shown to be true in a variety of bowel surgeries in adults. ICG has also been shown to be safe in children. Given that HD and ARM are both relatively rare conditions (~1/5000 live births), research in this area needs to be strategic. The investigators want to ensure that the investigators can recruit enough patients to the study using this protocol such that if this were to be scaled up to a multi-centre trial in the future, the investigators could demonstrate feasibility. The investigators will collect data both on the feasibility of recruitment as the primary outcome and secondary outcomes including stricture, leak, length of stay in hospital, and return to hospital.

DETAILED DESCRIPTION:
Pediatric colorectal conditions, such as Hirschsprung's disease (HD) and anorectal malformations (ARM), result in significant disease burden in pediatric populations in Canada. Both conditions are present in approximately 1 in 5000 live births. Surgical correction of these anomalies is typically performed in Children's Hospitals in Canada. Postoperative complications, such as anal stricture and anal stenosis, have been reported to occur in 2-35% and 2-10%, after posterior-sagittal anorectoplasty (PSARP) and laparoscopic-assisted pull through for ARM and HD, respectively. In addition, anastomotic leaks and dehiscence are life-threatening, and should be avoided at all costs. The literature estimates the rate of anastomotic leak in HD to be approximately 2%, but have been reported in as high as 10% in neonatal patients. Wound dehiscence post ARM repair has been estimated as high as 30-40%. It is hypothesized that the above post-operative complications occur due to compromised vascular supply to the bowel undergoing coloanal anastomosis at the time of pull-through.

Traditionally, surgeons evaluate bowel viability with tactile and visual means, including discoloration, bleeding from the cut edge, and peristalsis after resection. With the push towards minimally invasive surgeries over recent decades, the adoption of surgical technology which can replace open or tactile assessments is necessary. One such example is the use of indocyanine green (ICG) for assessing bowel perfusion in laparoscopic surgery. ICG is a nontoxic, nonimmunogenic, water-soluble intravascular imagine agent. It has a short half-life (approximately 3-5 minutes) and when injected intravenously, it binds to plasma proteins and proteins in the lymph fluid keeping it in the intravascular compartment. ICG absorbs light in the near-infrared region (806 nm) and emits fluorescent light at 830 nm. ICG was approved by the Food and Drug Administration (FDA, New Drug Application [NDA] 211580 505(b)(2) via fda.gov) for use in adults in the late 1950s and has since been approved for use in adults by Health Canada.

A review article published in 2012 identified over 200 manuscripts describing safe and reliable use of ICG in surgical procedures in adults. More specifically, qualitative analysis of bowel perfusion enhanced by ICG in colorectal cancer patients has been shown to reduce rates of anastomotic leak by approximately 4%. Practically speaking, the use of ICG florescence technique can be useful in identifying clinical vascular anatomy in colorectal surgery, both via open and laparoscopic approaches, allowing surgeons to better preserve important structures.

Several studies have shown that ICG is safe among pediatric populations, with utility demonstrated in cases of difficult cholecystectomy, hydrocele repairs, and localizing metastatic disease. As such, the FDA has approved the use of ICG in paediatric patients. Research studies from the US, have examined the intravenous application of ICG for more than 60 years in adults and children with few reported adverse effects. However, Health Canada has not reported on the safety and efficacy of ICG and does not authorize an indication for its use.

To our knowledge, there have only been two studies that have looked at intraoperative ICG to visualize intestinal perfusion for primary pull-through in Hirschsprung Disease and anorectal malformation repair patients and both were retrospective studies. A previous study included eight patients, diagnosed with HD undergoing transanal, open or laparoscopically-assisted pull-through procedures after biopsy confirmation of aganglionosis. Patients were given a dose of 1.25mg (<2 mg/kg) of ICG intraoperatively in the operating room. In five of the eight patients, the level of the bowel transection was changed based on the ICG visualization. In the other three patients, ICG confirmed the surgeon's assessment of where the resection should occur. There were no intraoperative complications or complications noted at two-week, one-month, and three-month follow-up visits. Further no leaks, incontinence, or strictures were noted at any of these follow-up visits. Another study 16 included 13 patients in total, nine undergoing cloacal reconstruction, four with HD and one with an ARM. ICG was used to predict the vascular supply during the reconstruction procedure and patients were given an intravenous dose of ICG between 0.1 to 0.3mg/kg in the operating room. There were no intraoperative adverse events or side effects from the ICG. ICG changed the operative plan in four out of 13 cases (31%), one of those four cases being a pull-through for HD. For this HD case, ICG resulted in the detection of 10cm of non-viable colon which may not have previously been detected. Although the level of evidence is limited by study design and small sample sizes, these studies help to provide rationale for the continued study of ICG use in paediatric patients.

Despite the results from these studies, future work is needed before he investigators can determine the effectiveness of ICG in reducing rates of post PSARP and pull-through complications. Practically speaking, the main inhibitors to widespread adoption of ICG in these surgeries is the cost of the technology, and lack of data to support that it truly reduces the rates of complications associated with these surgeries. Our research team, looks to be the first group to explore the feasibility of using ICG in a paediatric population with Hirschsprung's Disease and anorectal malformations. The investigators hope that the results from the study will help to initiate future multicenter, randomized controlled trials to provide high level evidence to support the use of ICG in colorectal surgeries in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with Hirschsprung's disease or anorectal malformations, diagnosed by:

   1. Clinical evaluation and physical examination
   2. Radiologic studies including abdominal x-rays and/or contrast enemas
   3. Pathologic diagnosis after rectal biopsies (HD only)
2. Patients greater than one-month of age to 7 years of age at the time of surgery
3. Patient requires surgical management for their diagnosis
4. Patient/Substitute decision maker (SDM) able to read/write/understand English

Exclusion Criteria:

1. Those patients and SDM unwilling to provide consent
2. Pregnant and/or women who are breast feeding
3. Patients with a known iodine allergy

Ages: 1 Month to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The number of eligible paediatric patients treated for HD or ARM at the local institute that would qualify for participation in this trial. | 12 months
  The number of eligible patients that are treated for HD and ARM at this institution regardless of if they enrolled in the study or not.
The number of eligible paediatric patients treated for HD or ARM that enroll in this study during the recruitment period of this study. | 12 months
  The number of eligible patient who enroll in this study during the recruitment period compared to the total number of eligible patient.
The number of eligible paediatric patients treated for HD or ARM that enroll in this study and attend al required study visits. | 12 months
  This outcome will capture the number of patient who are enrolled in the study and present to the hospital on the day of surgery, and for each follow-up visit where data will be collected.
The number of eligible paediatric patients treated for HD or ARM that enrolled in this study but are lost to attrition/drop-out during the study | 12 months
  This outcome captures the number of patient who enroll in the study but do not complete the study (including follow-up visits) or withdraw from the study before undergoing surgery.

SECONDARY OUTCOMES:
If the use of ICG alters the intraoperative management of the patient, resulting in the surgeon resecting a longer segment of bowel. | 5 hours
  This will be difference in where the surgeon would resect the bowel based on their clinical judgement and where the blood perfusion (indicated by ICG) suggests the resection should be made. This will be measure in millimeters.
If the use of ICG alters the length of operative time between ICG and control group | 5 hours
  This will be measured by comparing the length of operation for similar cases/diagnoses that are randomized to each study arm. This will be measured in minutes
If the use of ICG alters the length of stay in hospital between ICG and control group | 2 weeks
  This outcome will be tracked by measuring the length of hospital stay post-surgery for each patient enrolled in the study. This will be recorded in days.
Rates of anastomotic dehiscence | Up to 6 months post surgery
  This will be monitored as per standard surgical aftercare and monitoring by the surgeon. This data will be collected from the assessment of the surgeon and the patient's medical chart.
Rates of anal stricture (mild) not requiring anal dilatations | Up to 6 months post surgery
  This will be monitored as per standard surgical aftercare and monitoring by the surgeon. This data will be collected from the assessment of the surgeon and the patient's medical chart.
Rate of anal stricture (moderate or severe) requiring anal dilatations | Up to 6 months post surgery
  This will be monitored as per standard surgical aftercare and monitoring by the surgeon. This data will be collected from the assessment of the surgeon and the patient's medical chart.
Rate of hospital readmission in the first 30 days postoperatively | Up to 6 months post surgery
  This will be monitored as per standard surgical aftercare and monitoring by the surgeon. This data will be collected from the patient's medical chart.
Rate of an additional related procedure under general anaesthesia (i.e. return to the operating room or interventional radiology) | Up to 6 months post surgery
  This will be monitored as per standard surgical aftercare and monitoring by the surgeon. This data will be collected from the assessment of the surgeon and the patient's medical chart.

OTHER OUTCOMES:
Adverse reaction to ICG resulting in anaphylaxis | Up to 2 weeks post-op
  Patient will be monitored for this condition in the operating room during the surgery and up until they are discharged from hospital post-surgery.
Adverse reaction to ICG resulting in urticarial reactions | Up to 2 weeks post-op
  Patient will be monitored for this condition in the operating room during the surgery and up until they are discharged from hospital post-surgery.
Adverse reaction to ICG resulting in drug interactions | Up to 2 weeks post-op
  Patient will be monitored for this condition in the operating room during the surgery and up until they are discharged from hospital post-surgery.
Adverse reaction to ICG resulting in adverse events/complications | Up to 2 weeks post-op
  Patient will be monitored for this condition in the operating room during the surgery and up until they are discharged from hospital post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Butter, MD, Principal Investigator — Pediatric Surgeon, Children's Hospital, LHSC
Locations (1):
- Children's Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data (IPD)

REFERENCES:
- [Background] Mundt E, Bates MD. Genetics of Hirschsprung disease and anorectal malformations. Semin Pediatr Surg. 2010 May;19(2):107-17. doi: 10.1053/j.sempedsurg.2009.11.015. PMID 20307847
- [Background] Kudszus S, Roesel C, Schachtrupp A, Hoer JJ. Intraoperative laser fluorescence angiography in colorectal surgery: a noninvasive analysis to reduce the rate of anastomotic leakage. Langenbecks Arch Surg. 2010 Nov;395(8):1025-30. doi: 10.1007/s00423-010-0699-x. Epub 2010 Aug 12. PMID 20700603
- [Background] Tang ST, Wang GB, Cao GQ, Wang Y, Mao YZ, Li SW, Li S, Yang Y, Yang J, Yang L. 10 years of experience with laparoscopic-assisted endorectal Soave pull-through procedure for Hirschsprung's disease in China. J Laparoendosc Adv Surg Tech A. 2012 Apr;22(3):280-4. doi: 10.1089/lap.2011.0081. PMID 22449115
- [Background] Lu C, Hou G, Liu C, Geng Q, Xu X, Zhang J, Chen H, Tang W. Single-stage transanal endorectal pull-through procedure for correction of Hirschsprung disease in neonates and nonneonates: A multicenter study. J Pediatr Surg. 2017 Jul;52(7):1102-1107. doi: 10.1016/j.jpedsurg.2017.01.061. Epub 2017 Feb 2. PMID 28185631
- [Background] Engum SA, Grosfeld JL. Long-term results of treatment of Hirschsprung's disease. Semin Pediatr Surg. 2004 Nov;13(4):273-85. doi: 10.1053/j.sempedsurg.2004.10.015. PMID 15660321
- [Background] Ryu S, Suwa K, Kitagawa T, Aizawa M, Ushigome T, Okamoto T, Eto K, Yanaga K. Real-Time Fluorescence Vessel Navigation Using Indocyanine Green During Laparoscopic Colorectal Cancer Surgery. Anticancer Res. 2019 Jun;39(6):3009-3013. doi: 10.21873/anticanres.13433. PMID 31177142
- [Background] Elsaied A, Aly K, Thabet W, Magdy A. Two-stage repair of low anorectal malformations in girls: is it truly a setback?. Annals of Pediatric Surgery. 2013;9(2):69-73.
- [Background] Peng CH, Chen YJ, Pang WB, Zhang TC, Wang ZM, Wu DY, Wang K. STROBE-anastomotic leakage after pull-through procedure for Hirschsprung disease. Medicine (Baltimore). 2018 Nov;97(46):e13140. doi: 10.1097/MD.0000000000013140. PMID 30431584
- [Background] Tofft L, Salo M, Arnbjornsson E, Stenstrom P. Wound Dehiscence after Posterior Sagittal Anorectoplasty in Children with Anorectal Malformations. Biomed Res Int. 2018 Nov 11;2018:2930783. doi: 10.1155/2018/2930783. eCollection 2018. PMID 30534556
- [Background] Cassinotti E, Costa S, DE Pascale S, Oreggia B, Palazzini G, Boni L. How to reduce surgical complications in rectal cancer surgery using fluorescence techniques. Minerva Chir. 2018 Apr;73(2):210-216. doi: 10.23736/S0026-4733.18.07632-0. Epub 2018 Feb 21. PMID 29471617
- [Background] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Background] Wada T, Kawada K, Takahashi R, Yoshitomi M, Hida K, Hasegawa S, Sakai Y. ICG fluorescence imaging for quantitative evaluation of colonic perfusion in laparoscopic colorectal surgery. Surg Endosc. 2017 Oct;31(10):4184-4193. doi: 10.1007/s00464-017-5475-3. Epub 2017 Mar 9. PMID 28281123
- [Background] Esposito C, Del Conte F, Cerulo M, Gargiulo F, Izzo S, Esposito G, Spagnuolo MI, Escolino M. Clinical application and technical standardization of indocyanine green (ICG) fluorescence imaging in pediatric minimally invasive surgery. Pediatr Surg Int. 2019 Oct;35(10):1043-1050. doi: 10.1007/s00383-019-04519-9. Epub 2019 Jul 4. PMID 31273452
- [Background] Esposito C, Settimi A, Del Conte F, Cerulo M, Coppola V, Farina A, Crocetto F, Ricciardi E, Esposito G, Escolino M. Image-Guided Pediatric Surgery Using Indocyanine Green (ICG) Fluorescence in Laparoscopic and Robotic Surgery. Front Pediatr. 2020 Jun 17;8:314. doi: 10.3389/fped.2020.00314. eCollection 2020. PMID 32626676
- [Background] Rentea RM, Halleran DR, Ahmad H, Sanchez AV, Gasior AC, McCracken K, Hewitt GD, Alexander V, Smith C, Weaver L, Wood RJ, Levitt MA. Preliminary Use of Indocyanine Green Fluorescence Angiography and Value in Predicting the Vascular Supply of Tissues Needed to Perform Cloacal, Anorectal Malformation, and Hirschsprung Reconstructions. Eur J Pediatr Surg. 2020 Dec;30(6):505-511. doi: 10.1055/s-0039-1700548. Epub 2019 Dec 13. PMID 31858494
- [Background] Goldstein SD, Heaton TE, Bondoc A, Dasgupta R, Abdelhafeez A, Davidoff AM, Lautz TB. Evolving applications of fluorescence guided surgery in pediatric surgical oncology: A practical guide for surgeons. J Pediatr Surg. 2021 Feb;56(2):215-223. doi: 10.1016/j.jpedsurg.2020.10.013. Epub 2020 Oct 19. PMID 33189300
- [Background] Foppa C, Denoya PI, Tarta C, Bergamaschi R. Indocyanine green fluorescent dye during bowel surgery: are the blood supply "guessing days" over? Tech Coloproctol. 2014 Aug;18(8):753-8. doi: 10.1007/s10151-014-1130-3. Epub 2014 Feb 21. PMID 24558047
- [Background] Emran M, Wayne C, Koehler SM, Almond PS, Patel H. Intraoperative ICG-NIR Fluorescence Angiography Visualization of Intestinal Perfusion in Primary Pull-Through for Hirschsprung Disease. International Journal of Medical and Health Sciences. 2020 Nov 1;14(12):408-11
- [Background] Balamurugan S, Agrawal A, Kato Y, Sano H. Intra operative indocyanine green video-angiography in cerebrovascular surgery: An overview with review of literature. Asian J Neurosurg. 2011 Jul;6(2):88-93. doi: 10.4103/1793-5482.92168. PMID 22347330
- [Background] Cochran ST, Bomyea K, Sayre JW. Trends in adverse events after IV administration of contrast media. AJR Am J Roentgenol. 2001 Jun;176(6):1385-8. doi: 10.2214/ajr.176.6.1761385. PMID 11373197
- [Background] Hope-Ross M, Yannuzzi LA, Gragoudas ES, Guyer DR, Slakter JS, Sorenson JA, Krupsky S, Orlock DA, Puliafito CA. Adverse reactions due to indocyanine green. Ophthalmology. 1994 Mar;101(3):529-33. doi: 10.1016/s0161-6420(94)31303-0. PMID 8127574